CLINICAL TRIAL: NCT02594332
Title: A Randomized, Double-blind, Placebo-controlled, Mono-center Study to Evaluate the Effects of Mepolizumab on Airway Physiology in Patients With Eosinophilic Asthma: the MEMORY Study
Brief Title: Effects of Mepolizumab Compared to Placebo on Airway Physiology in Patients With Eosinophilic Asthma: MEMORY Study
Acronym: MEMORY
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: recruitment problems
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, PD Dr. Stephanie Korn, principal investigator, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-001; 2015-001868-19 (EudraCT Number)
Record Dates: First submitted 2015-08-31; First posted 2015-11-03 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Asthma
Keywords: eosinophilic asthma; mepolizumab; treatment
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia | interventions — mepolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mepolizumab (Experimental): 100 mg SC every 4 weeks for 13 injections
  Interventions: Drug: Mepolizumab
- Placebo (Experimental): Amount of Placebo corresponding to mepolizumab dose SC every 4 weeks for 13 injections
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mepolizumab — 100 mg SC every 4 weeks for 13 injections
  Arms: Mepolizumab
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the MEMORY trial is to compare the effects of mepolizumab with Placebo on airway physiology in patients with eosinophilic asthma

DETAILED DESCRIPTION:
Asthma with eosinophilic inflammation in the airways and/or blood eosinophilia is associated with clinical severity including the risk of exacerbations and relevant comorbidities (e.g. nasal polyposis). Interleukin-5 (IL-5) is a cytokine essential for eosinophil trafficking and survival. Clinical trials of blocking IL-5 with anti-IL-5 antibodies (mepolizumab and reslizumab) in patients with uncontrolled eosinophilic asthma resulted in an improvement in exacerbation rate and oral corticosteroid use. In some studies with mepolizumab and reslizumab there was a beneficial effect on lung function (FEV1). In addition, many patients described a profound impact on asthma symptoms and quality of life in personal reports which is not uniformly reflected in clinical trials.

The MEMORY trial is the first to primarily evaluate the effect of mepolizumab treatment on pulmonary function in patients with severe eosinophilic asthma. Importantly, using spirometry and bodyplethysmography will allow to evaluate additional parameters beyond FEV1 that more closely mirror the pathophysiological changes and functional aspects of airflow limitation in asthma in real life, e.g. airway resistance, hyperinflation and diffusion capacity. The proposed trial will answer the important questions: if, and if so, which parameters of airway (patho-) physiology as assessed by bodyplethysmography best reflect clinical response to mepolizumab therapy in patients with severe eosinophilic asthma. In addition, the time course to clinical response will be assessed. Equally important, there is only a loose correlation between FEV1 and parameters of asthma control and asthma-related quality of life. This is why another new and important aspect of this trial is to carefully monitor asthma control and asthma quality in life in correlation with lung function changes beyond FEV1. Finally, it is tempting to speculate that the proposed trial will contribute to the question how to best define clinical response to mepolizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be able to give written informed consent prior to participation in the study, which will include the ability to comply with the requirements and restrictions listed in the consent form.
2. Male or female patients at least 18 years
3. Physician-diagnosis of asthma and evidence of asthma as documented by either reversibility of airflow obstruction (FEV1 ≥ 12% or 200 ml) demonstrated at visit 1 or visit 2 .
4. ICS dose must be ≥ 1000 μg/day BDP or equivalent daily with or without maintenance oral corticosteroids.
5. Treatment in the past 12 months with an additional controller medication for at least 3 successive months, e.g., long-acting beta-2-agonist (LABA), leukotriene receptor antagonist (LTRA), or theophylline.
6. Persistent airflow obstruction as indicated by a pre-bronchodilator FEV1 < 80% predicted recorded at Visit 1 or < 90% for patients on oral corticosteroids.
7. An elevated peripheral blood eosinophil level of ≥ 300/µL that is related to asthma or ≥ 150/µL in patients treated with oral corticosteroids as maintenance therapy demonstrated at visit 1 or in the previous 12 months
8. Confirmed history of two or more exacerbations requiring treatment with systemic corticosteroids (intramuscular, intravenous, or oral), in the 12 months prior to visit 1, despite the use of high-dose inhaled corticosteroids. For patients receiving maintenance corticosteroids, the corticosteroid treatment for the exacerbations must have been a two-fold increase or greater in the dose.

Exclusion Criteria:

1. Current smokers or former smokers with a smoking history of ≥ 10 pack years (number of pack years = (number of cigarettes per day / 20) x number of years smoked). Patients who have not smoked for ≥ 6 months before visit 1 and have < 10 pack years can be included into the study.
2. Presence of a clinically important lung condition other than asthma. This includes current infection, bronchiectasis, pulmonary fibrosis, bronchopulmonary aspergillosis, or diagnoses of emphysema or chronic bronchitis (chronic obstructive pulmonary disease other than asthma) or a history of lung cancer.
3. Patients who have received omalizumab [Xolair] within 130 days of Visit 1.
4. Patients who have received any biological to treat inflammatory disease within 5 half-lives of visit 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-11-17 (Actual); Primary Completion 2017-05-22 (Actual); Study Completion 2017-05-22 (Actual)

PRIMARY OUTCOMES:
mean change from baseline in pre- and post-bronchodilator FVC at visit 10 (week 24) and at time of response | week 24 and time of response
  The primary outcome is the mean change from baseline in pre- and post-bronchodilator forced vital capacity (FVC) at visit 10 (week 24) and at time of response
mean change from baseline in pre- and post-bronchodilator FEV1 at visit 10 (week 24) and at time of response | week 24 and time of response
  The primary outcome is the mean change from baseline in pre- and post-bronchodilator forced expiratory volume in 1 second (FEV1) at visit 10 (week 24) and at time of response
mean change from baseline in pre- and post-bronchodilator RV at visit 10 (week 24) and at time of response | week 24 and time of response
  The primary outcome is the mean change from baseline in pre- and post-bronchodilator residual volume (RV) at visit 10 (week 24) and at time of response
mean change from baseline in pre- and post-bronchodilator TLC at visit 10 (week 24) and at time of response | week 24 and time of response
  The primary outcome is the mean change from baseline in pre- and post-bronchodilator total lung capacity (TLC) at visit 10 (week 24) and at time of response
mean change from baseline in pre- and post-bronchodilator airway resistance at visit 10 (week 24) and at time of response | week 24 and time of response
  The primary outcome is the mean change from baseline in pre- and post-bronchodilator airway resistance at visit 10 (week 24) and at time of response
mean change from baseline in pre- and post-bronchodilator IC at visit 10 (week 24) and at time of response | week 24 and time of response
  The primary outcome is the mean change from baseline in pre- and post-bronchodilator inspiratory capacity (IC) at visit 10 (week 24) and at time of response
mean change from baseline in pre- and post-bronchodilator CO diffusion capacity at visit 10 (week 24) and at time of response | week 24 and time of response
  The primary outcome is the mean change from baseline in pre- and post-bronchodilator CO diffusion capacity at visit 10 (week 24) and at time of response

SECONDARY OUTCOMES:
Mean change from baseline in pre- and post-bronchodilator forced vital capacity (FVC) over the 48-week treatment period at prespecified timepoints (1, 3, 6, 9 and 12 months) | 1, 3, 6, 9 and 12 months
Mean change from baseline in pre- and post-bronchodilator forced expiratory volume in 1 second (FEV1) over the 48-week treatment period at prespecified timepoints (1, 3, 6, 9 and 12 months) | 1, 3, 6, 9 and 12 months
Mean change from baseline in pre- and post-bronchodilator residual volume (RV) over the 48-week treatment period at prespecified timepoints (1, 3, 6, 9 and 12 months) | 1, 3, 6, 9 and 12 months
Mean change from baseline in pre- and post-bronchodilator total lung capacity (TLC) over the 48-week treatment period at prespecified timepoints (1, 3, 6, 9 and 12 months) | 1, 3, 6, 9 and 12 months
Mean change from baseline in pre- and post-bronchodilator airway resistance over the 48-week treatment period at prespecified timepoints (1, 3, 6, 9 and 12 months) | 1, 3, 6, 9 and 12 months
Mean change from baseline in pre- and post-bronchodilator inspiratory capacity (IC) over the 48-week treatment period at prespecified timepoints (1, 3, 6, 9 and 12 months) | 1, 3, 6, 9 and 12 months
Mean change from baseline in pre- and post-bronchodilator CO diffusion capacity over the 48-week treatment period at prespecified timepoints (1, 3, 6, 9 and 12 months) | 1, 3, 6, 9 and 12 months
Exercise tolerance in a subgroup of patients: Mean change from baseline in exercise endurance time | 1, 3, 6, 9 and 12 month
  Mean change from baseline in exercise endurance time during a sub-maximal constant-load cycle ergometry test after 1, 3, 6, 9 and 12 months of treatment.
Exercise tolerance in a subgroup of patients: Mean change from baseline in inspiratory capacity (IC) | 1, 3, 6, 9 and 12 month
  Mean change from baseline in inspiratory capacity (IC) at rest and at peak during sub-maximal constant-load cycle ergometry test after 1, 3, 6, 9 and 12 months of treatment.
Exercise tolerance in a subgroup of patients: Mean change from baseline in exertional dyspnea and leg discomfort (Borg CR10 Scale®) | 1, 3, 6, 9 and 12 month
  Mean change from baseline in exertional dyspnea and leg discomfort (Borg CR10 Scale®) during sub-maximal constant-load cycle ergometry test after 1, 3, 6, 9 and 12 months of treatment
Time to clinical response and time to change of baseline parameters of clinical Response: sence of smell | 52 weeks
Time to clinical response and time to change of baseline parameters of clinical Response: sense of taste | 52 weeks
Time to clinical response and time to change of baseline parameters of clinical Response: lung volume | 52 weeks
Time to clinical response and time to change of baseline parameters of clinical Response: CO Diffusion capacity | 52 weeks
Time to clinical response and time to change of baseline parameters of clinical Response: FEV1 reversibility | 52 weeks
Time to clinical response and time to change of baseline parameters of clinical Response: exhaled NO (eNO) | 52 weeks
Time to clinical response and time to change of baseline parameters of clinical Response: blood eosinophils | 52 weeks
Time to clinical response and time to change of baseline parameters of clinical Response: eosinophilic cationic Protein (ECP) | 52 weeks
Time to clinical response and time to change of baseline parameters of clinical Response: blood periostin | 52 weeks
Mean change from baseline in Asthma Control Questionnaire (ACQ) | 52 weeks
Mean change from baseline in Asthma Quality of Life Questionnaire (AQLQ) | 52 weeks
Mean change from baseline in St. George´s Respiratory Questionnaire (SQRG) | 52 weeks
Mean change from baseline in Dyspnoe Index (BDI/TDI) | 52 weeks
Mean change from baseline in fatique | 52 weeks
Mean change from baseline in number of days off school/work over the 48-week treatment period | 48 weeks
Time to first clinically significant exacerbation requiring oral or systemic corticosteroids, hospitalization, and/or emergency department (ED) visits | 52 weeks
Frequency of clinically significant exacerbations | 52 weeks
Time to first exacerbation requiring hospitalization or emergency department (ED) visit | 52 weeks
Frequency of exacerbations requiring hospitalization (including intubation and admittance to an intensive care unit (ICU)) or ED visits | 52 weeks
GETE rating by physician and patient at time of response and over the 52-week treatment period at pre-specified timepoints (1, 3, 6, 9 and 12 months) | 1, 3, 6, 9 and 12 month
Mean change in proportion of patients with nasal polyps, chronic sinusitis and loss of smell and taste | 52 weeks
Clinical response to mepolizumab in relation to asthma parameters which potentially predict clinical response | 52 weeks
  Clinical response to mepolizumab in relation to asthma parameters which potentially predict clinical response (age at onset and duration of asthma, prior asthma medication, presence of nasal polyps, sense of smell and taste, allergic sensitization (skin prick test, total and specific IgE against aeroallergens and Staph. aureus enterotoxin), reversibility of airflow obstruction, eNO, blood eosinophils, eosinophilic cationic protein (ECP), blood periostin, ANA, ANCA, ECP.
Routine safety assessment (AE and SAE reporting, withdrawals, pregnancy, hematological and clinical chemistry parameters, ECG and vital signs (pulse rate and systolic and diastolic blood pressure)) | 52 weeks
  Routine safety assessments are incorporated throughout and/or at the end of treatment period including AE and SAE reporting, withdrawals, pregnancy, hematological and clinical chemistry parameters, ECG and vital signs (pulse rate and systolic and diastolic blood pressure).

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Korn, MD, Principal Investigator — Johannes Gutenberg University Mainz
Locations (1):
- Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Pneumologie, Mainz, Germany

IPD SHARING:
Plan to Share IPD: Undecided